CLINICAL TRIAL: NCT00498290
Title: The Protocol of Enhanced Recovery After Surgery in Colorectal Surgery
Acronym: ERAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: xu jianmin, department of general surgery, zhongshan hospital, fudan university
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-51
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Colorectal Surgery
Keywords: Enhanced Recovery After Surgery Protocol(ERAS); Colorectal Surgery
MeSH Terms: interventions — Enhanced Recovery After Surgery; Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): received enhanced recovery after surgery (ERAS) protocol in colorectal surgery
  Interventions: Procedure: enhanced recovery after surgery (ERAS) protocol
- B (No Intervention): normal recovery protocol in colorectal surgery
  Interventions: Procedure: control

INTERVENTIONS:
Procedure: enhanced recovery after surgery (ERAS) protocol — An integrated protocol aims to allow patients to recover more quickly from major surgery, avoid medium-term sequelae of conventional postoperative care (e.g. decline in nutritional status and fatigue) and reduce health care costs by reducing hospital stay
  Arms: A
Procedure: control — normal recovery protocol as usually
  Arms: B

SUMMARY:
The purpose of this study is to determine whether ERAS is safe and can decrease surgical stress, increase functional recovery and reduce complication rate in colorectal surgery.

DETAILED DESCRIPTION:
The key factors that keep a patient in hospital after uncomplicated major colorectal surgery include the need for parenteral analgesia(persistent pain), intravenous fluids (persistent gut dysfunction), and bed rest (persistent lack of mobility). These factors often overlap and interact to delay return of function. Obviously, postoperative complications will also prolong the time until recovery and ultimately length of stay. A clinical pathway, called Enhanced Recovery After Surgery(ERAS), to accelerate recovery after colonic resection based on a multimodal programme with optimal pain relief, stress reduction with regional anaesthesia, early enteral nutrition and early mobilisation has demonstrated improvements in physical performance, pulmonary function, body composition and a marked reduction of length of stay.

Comparison(s): A total of 500 cases colorectal surgery were randomized to receive ERAS protocol or the traditional protocol, such as mechanical bowl preparation, intravenous fluids until bowl movement recovery and bed rest.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal surgery patients
* Age 20～80
* Without comorbidities which will influence prognosis, such as paralysis, spine cataface, or cardiac infarction

Exclusion Criteria:

* Emergency
* Combined other organ resection
* Age > 80
* Comorbidities which will influence prognosis, such as paralysis, spine cataface, or cardiac infarction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
safety of the ERAS protocol and whether it can decrease surgical stress, increase functional recovery and reduce complication rate in colorectal surgery | perioperation and until 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: jianmin xu, professor, Study Chair — department of general surgery, zhongshan hospital, fudan university
Locations (1):
- Department of General Surgery, Zhongshan Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Derived] Ren L, Zhu D, Wei Y, Pan X, Liang L, Xu J, Zhong Y, Xue Z, Jin L, Zhan S, Niu W, Qin X, Wu Z, Wu Z. Enhanced Recovery After Surgery (ERAS) program attenuates stress and accelerates recovery in patients after radical resection for colorectal cancer: a prospective randomized controlled trial. World J Surg. 2012 Feb;36(2):407-14. doi: 10.1007/s00268-011-1348-4. PMID 22102090